CLINICAL TRIAL: NCT07393074
Title: Involvement of the Autonomic Nervous System in Hepatocellular Carcinoma (HCC): a Pilot Psycho-behavioral and Neurophysiological Study
Brief Title: PSYLIVER-PILOTE: Involvement of the Autonomic Nervous System in Hepatocellular Carcinoma (HCC)
Acronym: PSYLIVER-PILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL25_0750; 2025-A01879-40 (Other: ID-RCB)
Record Dates: First submitted 2026-01-13; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hepato Cellular Carcinoma; Cirrhosis; Autonomic Nervous System; Central Nervous System
Keywords: HCC; cirrhosis; ANS; NRS
MeSH Terms: conditions — Fibrosis | interventions — epicatechin gallate

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, case-control pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with histologically proven cirrhosis based on liver biopsy performed as part of routine car (Experimental): * Information gathering: patient history, medical history and current treatments, clinical examination and available paraclinical tests, assessment of alcohol consumption
  * A dedicated consultation at the Croix Rousse hospital to perform:
    * Measurements of autonomic nervous system (ANS) activity at rest and during sensory stimulation.
    * Self-administered questionnaires to assess psycho-behavioral traits
  * Analysis of nocturnal cardiac activity (at home): electrocardiographic (ECG) recording of heart activity during one night.
  * A study of the liver biopsy (performed as part of routine care) will be carried out to analyze ANS activity at the intrahepatic level for calculating the NRS score
  Interventions: Other: Measurements of autonomic nervous system (ANS) activity at rest and during sensory stimulation.; Other: Self-administered questionnaires to assess psycho-behavioral traits; Other: Analysis of nocturnal cardiac activity (at home): electrocardiographic (ECG) recording of heart activity during one night.; Other: Calculation of the NRS score. A study of the liver biopsy will be carried out to analyze ANS activity at the intrahepatic level.; Other: Intervention name 5 * (Limit: 100 characters) Optionnal biocollection
- Patients with cirrhosis complicated by HCC, histologically confirmed by liver biopsy performed as pa (Experimental): * Information gathering: patient history, medical history and current treatments, clinical examination and available paraclinical tests, assessment of alcohol consumption
  * A dedicated consultation at the Croix Rousse hospital to perform:
    * Measurements of autonomic nervous system (ANS) activity at rest and during sensory stimulation.
    * Self-administered questionnaires to assess psycho-behavioral traits
  * Analysis of nocturnal cardiac activity (at home): electrocardiographic (ECG) recording of heart activity during one night.
  * A study of the liver biopsy (performed as part of routine care) will be carried out to analyze ANS activity at the intrahepatic level for calculating the NRS score
  Interventions: Other: Measurements of autonomic nervous system (ANS) activity at rest and during sensory stimulation.; Other: Self-administered questionnaires to assess psycho-behavioral traits; Other: Analysis of nocturnal cardiac activity (at home): electrocardiographic (ECG) recording of heart activity during one night.; Other: Calculation of the NRS score. A study of the liver biopsy will be carried out to analyze ANS activity at the intrahepatic level.; Other: Intervention name 5 * (Limit: 100 characters) Optionnal biocollection

INTERVENTIONS:
Other: Measurements of autonomic nervous system (ANS) activity at rest and during sensory stimulation. — Participants are informed that they will need to watch the screen, on which images will appear around a central symbol. They must click the mouse button as quickly as possible when they see an "x" sign and do nothing when they see a "+" sign appear in the center of the screen.
  Sensory stimulation is carried out using OpenSesame software. It is divided into four blocks of seven minutes each, with a break systematically offered to participants between each block. Each block comprises three phases: rest (sitting with hands on knees, palms facing upwards and eyes closed) for two minutes, responding to stimuli according to instructions for three minutes, and a second rest phase for two minutes. In fact, participants are only active for a total of 12 minutes. The blocks are presented in the same order for all participants: Go block, neutral Go/NoGo block, emotional Go/NoGo block, then social Go/NoGo block.
Other: Self-administered questionnaires to assess psycho-behavioral traits — Participants answer self-questionnaires on tablets by selecting the answer that seems most appropriate to them. They are told that there are no right or wrong answers and that they should answer as honestly as possible based on what they think and feel at that moment. The self-questionnaires are the QA-10 items, the short version of the UPPS-P, the BPAQ-SF, the CERQ, the DEX, the PSS-10, the HAD, and the ISI.
Other: Analysis of nocturnal cardiac activity (at home): electrocardiographic (ECG) recording of heart activity during one night. — The investigator presents the NeuroCoach test kit to the participant and gives it to them. This kit consists of a recorder, two electrodes, a single-use pouch for nighttime use, a prepaid envelope for returning the equipment, and installation instructions. The investigator explains the installation instructions for the device, which the participant will set up independently at home.
  The equipment used is CE 60601-1 certified (general requirements for basic safety and essential performance of medical electrical equipment). There is a risk of temporary local skin irritation where the electrodes come into contact with the skin.
  A prepaid envelope will be given to the patient to return the device.
Other: Calculation of the NRS score. A study of the liver biopsy will be carried out to analyze ANS activity at the intrahepatic level. — Liver biopsy is performed as part of routine care. After pathological analysis as part of routine care, the biopsy sample will be sent to the Unité PaThLiv laboratory (UMR UCBL1 INSERM U1350; PathLiv team) for NRS histological scoring.
Other: Intervention name 5 * (Limit: 100 characters) Optionnal biocollection — Venous blood samples (taken during two visits): for a total volume of 32mL(serum, plasma) for the biobank will be aliquoted and stored in cryotubes. Each sample taken will be labeled with the patient's anonymized code (the patient's first and last names will not appear on the tubes). The tubes will be transported to the laboratory (PaThLiv Unit - UMR UCBL1 INSERM U1350; PathLiv Team).

SUMMARY:
Chronic liver diseases affect 1.5 billion people worldwide and can lead to cirrhosis and hepatocellular carcinoma (HCC), which ranks as the third leading cause of cancer-related mortality globally. Despite advances in the treatment of hepatitis B and C, metabolic diseases, and addiction, HCC incidence continues to rise. In France, between 2010 and 2015, the five-year survival rate for liver cancer (90% of which is HCC) was 18% for men and 19% for women. Treatment of HCC is based on the BCLC classification (Barcelona Clinic Liver Cancer), which evaluates both cancer progression and liver function (Child-Pugh classification). Patients at early stages (0 or A) have a survival rate of over 5 years, while those at more advanced stages (C or D) have significantly lower survival rates, highlighting the importance of better early detection tools.

Current screening for HCC in cirrhotic patients involves biannual US-scan. However, ultrasound sensitivity for detecting tumors smaller than 2 cm is around 25%. Therefore, developing personalized strategies to predict and detect early-stage HCC is crucial to improving patient outcomes. Various clinical and biological scores have been developed to assess the risk of developing HCC in cirrhotic patients, but these scores remain imperfect. Molecular heterogeneity in HCC, as revealed by transcriptomic studies, could explain the variability in outcomes and treatment responses. This heterogeneity in occurrence, phenotype, and progression of HCC suggests individual singularities that are not yet well understood.

These individual singularities are likely linked to the autonomic nervous system (ANS), particularly in the central nervous system (CNS), which regulates various physiological processes. The ANS consists of the sympathetic nervous system (SNS), mainly adrenergic, and the parasympathetic nervous system (PNS), mainly cholinergic. These two systems function antagonistically but with different temporal dynamics. A better understanding of the interaction between tumor cells and their environment through the ANS could lead to the identification of new biomarkers to predict HCC development and therapeutic targets.

The role of the ANS in cancer development has been explored in various cancers, including prostate, stomach, pancreatic, breast, and ovarian cancers, where the ANS regulates inflammation and immune responses. In chronic liver diseases, the liver is innervated by both sympathetic and parasympathetic fibers, and this innervation plays a role in regulating metabolism, liver regeneration, and fibrosis progression. Chronic liver disease etiologies, such as alcohol consumption, metabolic syndrome, and viral hepatitis, disrupt the balance between the SNS and PNS, contributing to liver dysfunction. The severity of liver damage is linked to autonomic dysfunction, and heart rate variability, a marker of PNS activity, is correlated with survival in patients with terminal-stage HCC.

Our recent research has shown that patients with HCC exhibit a reconfiguration of the intrahepatic ANS, with a consistent cholinergic orientation at the neuro-hepatic synapse. Patients with parasympathetic orientation (as compared to sympathetic orientation) have more aggressive tumors, shorter survival, and, from a pharmacological perspective, anticholinergics increase sensitivity to targeted HCC therapies. Tumor cells and cytotoxic lymphocytes are most strongly associated with cholinergic receptor enrichment and depletion, respectively.

In this context, the PSYLIVER-PILOTE study builds on these findings by investigating the involvement of the ANS in HCC through non-invasive extra-hepatic measures. The SNS and PNS are connected to brain regions involved in cognitive, emotional, and social information processing, such as the anterior cingulate cortex, insula, ventromedial prefrontal cortex, amygdala, and hypothalamus. These brain areas are involved in cognitive control and emotional processing. Additionally, experimental data from polyvagal theory and neurovisceral integration theory highlight the role of the ANS in regulating cognitive, emotional, and social processes, as well as psycho-behavioral traits. For instance, confronting a person with cognitive tasks and emotional or social information alters the balance of sympathetic and parasympathetic activity. Similar changes are observed in psycho-behavioral disorders like depression, emotional dysregulation, stress, and aggression.

Thus, the PSYLIVER-PILOTE study aims to identify extra-hepatic markers of ANS activity associated with HCC, analyzing both electrophysiological indices (from the peripheral nervous system) and psycho-behavioral indices (from the central nervous system). This project could open new avenues for early HCC detection and the development of personalized treatments

ELIGIBILITY:
Inclusion Criteria:

Group A:

* Over 18 years of age
* Affiliated with a social security system
* Sufficient command of the French language to hold a conversation and read
* Signature of an informed consent form
* Compensated cirrhosis classified as CHILD-Pugh A with clinical indication for liver biopsy (either for the etiological diagnosis or confirmation of cirrhosis, or for the etiological diagnosis of liver damage)
* Liver biopsy scheduled as part of routine care for a diagnosis of cirrhosis without HCC

Group B:

* Over 18 years of age
* Affiliated with a social security system
* Sufficient command of the French language to hold a conversation and read
* Signature of an informed consent form
* Compensated cirrhosis classified as CHILD-Pugh A with clinical indication for liver biopsy (either for the etiological diagnosis of cirrhosis or its confirmation; or for the etiological diagnosis of liver damage)
* Liver biopsy scheduled as part of routine care for the diagnosis of suspected HCC (based on standard imaging criteria)

Exclusion Criteria:

* Personal history of cancer in the broad sense (including HCC prior to inclusion in the study)
* Pregnant or breastfeeding women
* Adults subject to legal protection measures (guardianship, curatorship)
* Contraindications to trans-parietal liver biopsy: clinical or radiological ascites, coagulation disorders, curative anticoagulation that cannot be suspended, dilation of the bile ducts
* Persons deprived of their liberty by judicial or administrative decision
* Wearers of electronic implants (pacemakers, implantable cardioverter defibrillators, cochlear implants, brain implants, etc.)
* Psychotic disorders
* Degenerative neurological disorders (Parkinson's disease and related disorders, dementia, Korsakoff's syndrome, etc.)
* Antiarrhythmic treatment:

  * Class Ia: Disopyramide and Quinidine
  * Class Ic: Flecainide and Propafenone
* Neuroleptic psychotropic treatment affecting the ANS (haloperidol, chlorpromazine, olanzapine, clozapine, quetiapine), tricyclic antidepressants (e.g., amitriptyline, amoxapine, clomipramine, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
RNA expression values encoding all adrenergic receptors, and all cholinergic receptors or subunits. | At liver biopsy, within 6 months after inclusion
  The NRS is based on the RNA expression values of 6 human genes encoding all adrenergic receptors, and 21 genes encoding all cholinergic receptors or subunits.
  The NRS is defined by the difference between the sum of the expression values of adrenergic receptors on the one hand, and the sum of the expression values of cholinergic receptors on the other hand. Hence, the lower the NRS, the more cholinergic the sample is.

SECONDARY OUTCOMES:
Identify autistic traits | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A short screening questionnaire (AQ-10 (Autism Spectrum Quotient - 10 items)) designed to identify autistic traits in adults, focusing on social skills, attention switching, communication, and imagination.
Measure assessing five dimensions of impulsivity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A self-report measure assessing five dimensions of impulsivity: negative urgency, positive urgency, lack of premeditation, lack of perseverance, and sensation seeking.
Measure assessing different aspects of aggression | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A questionnaire (BPAQ (Buss-Perry Aggression Questionnaire)) measuring different aspects of aggression, including physical aggression, verbal aggression, anger, and hostility.
Evaluation of the cognitive strategies individuals | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A self-report instrument (CERQ (Cognitive Emotion Regulation Questionnaire)) that evaluates the cognitive strategies individuals use to regulate their emotions after experiencing stressful or negative events.
Measure assessing everyday problems related to executive dysfunction | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A measure (DEX (Dysexecutive Questionnaire)) assessing everyday problems related to executive dysfunction, such as difficulties with planning, emotional regulation, inhibition, and self-awareness.
Screening to detect symptoms of anxiety and depression | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A screening tool (HADS (Hospital Anxiety and Depression Scale)) designed to detect symptoms of anxiety and depression, particularly in medical or clinical settings, while minimizing the influence of physical symptoms.
Measure of heart rate variability | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion
  A global measure of heart rate variability (SDNN (Standard Deviation of NN intervals)) reflecting overall autonomic nervous system activity.
An index of parasympathetic (vagal) activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion
  An index (pNN50 (Percentage of NN intervals differing by more than 50 ms) of parasympathetic (vagal) activity based on short-term heart rate variability.
Measure of HRV reflecting parasympathetic nervous system activity. | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A time-domain (rMSSD (Root Mean Square of Successive Differences)) measure of HRV mainly reflecting parasympathetic nervous system activity.
Measure of total variance of heart rate variability | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  The total (Ptot (Total Power)) variance of heart rate variability across all frequency bands, reflecting overall autonomic regulation.
An index (HF (High-Frequency)) of the parasympathetic activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  An index of the parasympathetic activity .
An index often used to estimate the balance between sympathetic and parasympathetic activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  An index (LF/HF-HRV Ratio) often used to estimate the balance between sympathetic and parasympathetic activity (with interpretative limitations).
A measure of cardiac vagal modulation. | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A measure (DC (Deceleration Capacity)) of the heart's ability to slow down, reflecting cardiac vagal modulation.
Mesure spectrale du pouls cardiaque | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A spectral measure (PIP (Pulse Interval Power)) of pulse interval variability indicating autonomic modulation of heart rate.
A measure associated with slow regulatory mechanisms of the autonomic nervous system | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A measure (VLFI (Very Low Frequency Index)) associated with slow regulatory mechanisms of the autonomic nervous system, including thermoregulation and hormonal influences.
A measure of rapid changes in skin conductance | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A measure (EDR (Electrodermal Response)) of rapid changes in skin conductance reflecting phasic sympathetic nervous system activity.
A tonic measure of skin conductance | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A tonic measure of skin conductance (SCL (Skin Conductance Level)) indicating baseline sympathetic arousal.
A cardiac measure inversely related to sympathetic activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A cardiac measure inversely (PEP (Pre-Ejection Period)) related to sympathetic activity; shorter PEP reflects increased sympathetic drive.
A frequency-domain measure associated with parasympathetic (vagal) activity and respiratory influences. | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A frequency-domain measure (HF-HRV (High-Frequency Heart Rate Variability)) associated with parasympathetic (vagal) activity and respiratory influences.
An index representing overall sympathetic nervous system activation | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A composite index (SAI (Sympathetic Activity Index)) representing overall sympathetic nervous system activation.
An index representing overall parasympathetic (vagal) nervous system activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A composite index (PAI (Parasympathetic Activity Index)) representing overall parasympathetic (vagal) nervous system activity.
An index describing the relative balance between sympathetic and parasympathetic cardiac control | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion
  An index (CAB (Cardiac Autonomic Balance)) describing the relative balance between sympathetic and parasympathetic cardiac control
Measure the contribution of sympathetic activity to cardiac autonomic regulation | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion
  A measure (CSAB (Cardiac Sympathetic Autonomic Balance)) emphasizing the contribution of sympathetic activity to cardiac autonomic regulation.
An indicator of overall effectiveness and flexibility of autonomic control over cardiac function | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion
  An indicator (CAR (Cardiac Autonomic Regulation)) of overall effectiveness and flexibility of autonomic control over cardiac function.
Measure reflecting the efficiency of sympathetic regulation of cardiac activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion
  A measure (CSAR (Cardiac Sympathetic Autonomic Regulation)) reflecting the efficiency of sympathetic regulation of cardiac activity
A ratio expressing dominance of sympathetic versus parasympathetic autonomic activity | During the visit, before the liver biopsy, within a maximum of 6 months after inclusion.
  A ratio (SAI/PAI Ratio) expressing the relative dominance of sympathetic versus parasympathetic autonomic activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France